CLINICAL TRIAL: NCT04210336
Title: Estudio clínico, Aleatorizado, Doble Ciego, Paralelo, Controlado Con Gel de ácido láctico Para Evaluar la Eficacia Del Gel Papilocare® en la reparación de Lesiones Cervicales Causadas Por VPH. A Randomized, Double-blind, Parallel-group, Controlled Clinical Trial Using Lactic Acid Gel to Evaluate the Efficacy of Papilocare® Gel in Repairing Cervical Lesions Caused by HPV.
Brief Title: Clinical Trial to Evaluate Papilocare® Gel Efficacy Into Repairment of Cervical Lesions Caused by HPV
Acronym: PAPILOCAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Procare Health Iberia S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PAPILOCAN
Record Dates: First submitted 2019-12-11; First posted 2019-12-24 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: HPV Infection; Lesion Cervix
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PAPILOCARE (Experimental): Randomized patients will receive two different guidelines depending on the time of randomization:
  * Guideline A (from patient 1 to 100 in order of randomization): guideline of 1 cannula per day x 21 days + 7 days rest during the 1st month + 1 cannula / alternate days until completing 6 months (except for menstruation days ).
  * Guideline B (from patient 101 to 200 in order of randomization): pattern of 1 cannula per day x 21 days + 7 days rest for 3 months + 1 cannula / alternate days until completing 6 months (except for menstruation days) .
  Interventions: Device: PAPILOCARE
- LACTIC ACID GEL (Active Comparator): Randomized patients will receive two different guidelines depending on the time of randomization:
  * Guideline A (from patient 1 to 100 in order of randomization): guideline of 1 cannula per day x 21 days + 7 days rest during the 1st month + 1 cannula / alternate days until completing 6 months (except for menstruation days ).
  * Guideline B (from patient 101 to 200 in order of randomization): pattern of 1 cannula per day x 21 days + 7 days rest for 3 months + 1 cannula / alternate days until completing 6 months (except for menstruation days) .
  Interventions: Device: LACTIC ACID GEL

INTERVENTIONS:
Device: PAPILOCARE — Papilocare®: Vaginal Gel based on Coriolus versicolor, medical device class IIa.
  Route of administration: topical (vaginal). Papilocare® consists of the following ingredients: hyaluronic acid niosomes, β-glucans (magnolol, honokiol and carboxymethyl betaglucan) niosomes, BioEcolia® (Alpha-oligoglycan), Coriolus versicolor, Azadirachta indica (Neem) extract, Centella asiatica and Aloe vera.
  Arms: PAPILOCARE
Device: LACTIC ACID GEL — The lactic acid gel consists of a carrier gel with the absence of the active ingredients of Papilocare®.
  Arms: LACTIC ACID GEL

SUMMARY:
Clinical Trial phase III, randomized, double-blind, parallel-group, controlled using lactic acid gel to evaluate the efficacy of Papilocare gel in the repair of cervical lesions caused by HPV.

The study is divided into two parts. All patients included in the study will be randomized (1: 1) to one of the 2 study groups, Papilocare or lactic acid gel, using a randomization list and in double-blind conditions.

DETAILED DESCRIPTION:
Phase III, randomized, double-blind, parallel-group, controlled using lactic acid gel clinical trial to evaluate the efficacy of Papilocare gel in the repair of cervical lesions caused by HPV.

The study is divided into two parts. All patients included in the study will be randomized (1: 1) to one of the 2 study groups, Papilocare or lactic acid gel, using a randomization list and in double-blind conditions.

The study is divided into 2 parts, the first 100 randomized patients will receive treatment with an administration regimen in both arms: 1 cannula / day for 1 month + 1 cannula on alternate days for 5 months (except for menstruation days). The second part of the study, randomized patients from position 101 to 200, will receive treatment with an administration regimen in both arms: 1 cannula / day for 3 months + 1 cannula on alternate days for 3 months (except the days of menstruation).

Duration of treatment: 6 months Total study duration: 13 months in 5 visits: selection visit, V0 or randomization visit (30 days), V1(Month 3), V2 (Month 6), V3 (Month 12).

ELIGIBILITY:
Inclusion Criteria:

1. Woman between the ages of 30 and 65 (both included).
2. Able to read and understand the Patient Information Sheet and informed consent
3. Accept participation in the study and sign the Informed Consent.
4. Cytological result of ASC-US or LSIL, with concordant colposcopic image, at most 3 months before the selection visit. It is considered concordant with ASCUS and LSIL, a colposcopic result of normality, of non-specific findings or of type 1 changes.
5. Positive HPV according to cobas 4800 technique (high-risk HPV) carried out in a selection visit (or positive available at most 3 months prior to the baseline visit).
6. Women vaccinated and not vaccinated against HPV.
7. Is able, at the discretion of the researcher, to comply with the requirements of the study and without impediments to follow the instructions and assessments throughout it.

Exclusion Criteria:

1. Clinically relevant alterations of the immune system or any other autoimmune disease or in treatment with immunosuppressants.
2. Other cytological results other than those provided for in the inclusion criteria.
3. Baseline LSIL biopsies with CIN-3.
4. Abnormal undiagnosed genital bleeding (during the 6 months prior to the selection visit)
5. Other symptomatic vulvovaginal infections.
6. Surgical cervical excision in the last year or total hysterectomy.
7. Previous history of gynecological cancer.
8. Participation in any other clinical trial at present or in the 4 weeks prior to inclusion of the study.
9. Any planned surgery that precludes correct compliance with the guideline.
10. Use of vaginal contraceptives or other vaginal hormonal treatments.
11. Contraindications to the use of Papilocare® gel or known allergies to any of its components.
12. Women of childbearing age who do not use effective contraceptive methods, pregnant women, with suspected pregnancy or breastfeeding.

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-08-07 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
cervical mucosal repair | 6 months
  Percentage of patients with cervical lesions negativization confirmed be cytology and accordance colposcopy , at 6 months will be used to evaluate the main variables, degree of cervical mucosal repair in HPV-positive women with ASC-US or LSIL.

SECONDARY OUTCOMES:
Reepithelialization degree of the cervical mucosa | at 3 months
  Percentage of patients with negativity of cervical lesions by cytology and accordance colposcopy, at 3 months
Percentage of patients with Viral clearance | 3 and 6 months.
  Percentage of patients with initial HPV clearance measured by PCR at 3 and 6 months.
Vaginal health status measured by vaginal health index (VHI) | 3 and 6 months.
  Changes in the VHI (vaginal health index -Bachmann) at 3 and 6 months.
  VHI was developed in order to objectively assess female urogenital health (Bachmann GMaturitas. 1995 Dec; 22 Suppl():S1-S5.). This test evaluates overall elasticity, fluid secretion type and consistency, vaginal pH, epithelial mucosa and moisture. Minimum score is 5 and maximum is 25. Lower scores corresponds to greater urogenital atrophy.
Stress perceived by patients measured by PSS-14 (Perceived Stress Scale 14 items) | 3 and 6 months.
  Changes PSS-14 scale (Perceived Stress Scale 14 items) at 3 and 6 months.
  The PSS-14 is comprised of 14 items, score ranges from 0-56, with higher scores indicating greater perceived stress
Safety and tolerability of Papilocare® gel: Record of the incidence, nature and severity of adverse events | 6 months
  Record of the incidence, nature and severity of adverse events: during the 6 months of treatment duration.
Satisfaction degree with Papilocare gel use: Likert type scale | 3 and 6 months.
  Patients satisfaction degree with papilocare gel use as treatment will be evaluated by a likert type scale.
  A Likert scale is a psychometric scale commonly involved in research that employs questionnaires. It is the most widely used approach to scaling responses in survey research.Likert scaling assumes distances between each choice (answer option) are equal. Higher scores corresponds to better satisfaction with papilocare gel use.

OTHER OUTCOMES:
Change of biopsy results (optional) | 3 and 6 months.
  Only in cases that a biopsy has been performed per routine, the change or maintenance of biopsy results will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Alfonso Quesada López-Fe, Doctor, Principal Investigator — H Nuestra Señora de la Candelaria
Locations (1):
- Hospital Universitario Nuestra Señora de la Candelaria, Santa Cruz de Tenerife, Tenerife, Spain

IPD SHARING:
Plan to Share IPD: Yes
The PI from the participant site received the study protocol and the informed consent form previously to the initiation of the study and every time it occurs an amendment over the protocol, ICF or any other study document. Once the study will finish and the data will be analyzed, the PI will receive the CSR.
Supporting Information: Study Protocol, ICF, CSR